CLINICAL TRIAL: NCT06365593
Title: A Multicenter Observational retrosPective Registry of patIents With Transthyretin aMyloid polynEuropathy (hATTR-PN) and chRonic Idiopathic Axonal Polyneuropathy (CIAP) in the Population of the Russian Federation
Brief Title: hATTR Polyneuropathy in Russia
Acronym: PRIMER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8450R00005
Record Dates: First submitted 2024-03-01; First posted 2024-04-15 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hereditary Transthyretin Amyloidosis
Keywords: hATTR; CIAP; hATTR-PN; ATTR-PN; ATTRv; ATTR; polyneuropathy; transthyretin amyloid polyneuropathy; chronic idiopathic axonal polyneuropathy; hereditary transthyretin amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Polyneuropathies; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Patients with hATTR-PN: 50 adult patients with hATTR-PN
- Patients with CIAP: 50 adult patients with CIAP

SUMMARY:
A multicenter observational retrosPective Registry of patIents with transthyretin aMyloid polynEuropathy (hATTR-PN) and chRonic idiopathic axonal polyneuropathy (CIAP) in the population of the Russian Federation (PRIMER) There are no comprehensive epidemiological data on patients with hereditary ATTR-PN (hATTR-PN) and CIAP in the Russian Federation. Therefore, there is a need to conduct a large-scale observational study in the Russian population to obtain information on clinical, electrophysiological and demographic characteristics of patients with hATTR-PN and CIAP. Obtaining the study data will help to identify the patients with axonal polyneuropathy, who deserve TTR gene sequencing, and therefore to allow early treatment and potentially modify disease progression in patients.

DETAILED DESCRIPTION:
Since the increasing number of treatments available to help slow the progression of neuropathy it is critical to timely identify and diagnose the ATTR-PN. Early identification and intervention are also crucial to improve patient outcomes because newly available treatments have been shown to have maximum therapeutic benefit when started in the early stages of the disease.

Identification of ATTRv amyloidosis with PN can be challenging, particularly in non-endemic regions, and a high level of suspicion is required to diagnose patients as early as possible.

Previously proposed suspicion index of ATTRv amyloidosis was based on disease's red flags, that is, on the presence of a progressive polyneuropathy in addition to at least one red flag symptom suggestive of multi-systemic involvement. However, sometimes the demonstration of a progressive neuropathy requires follow-up evaluations, risking wasting time. Moreover, some red flags (e.g., cardiomyopathy or vitreous opacities) need specialist evaluations that could be often lacking during the first neurological evaluation.

Patients can present with heterogeneous symptoms and variable levels of disease severity, which often leads to a misdiagnosis. Early and accurate diagnosis may also be confounded by a lack of family history and the presence of various phenotypes common to multiple disease conditions such as GI disorders. In fact, CIAP still represents a common misdiagnosis for ATTRv patients.

Study is planned to determine the principal differences between the hATTR-PN and CIAP patients and valorize them in a compound score which can help clinician through a specific cut-off to recognize patients deserving TTR genetic analysis. The application of the compound score in patients with sensory-motor neuropathy may have a major role, representing a screening tool to avoiding wasting time and therefore shortening the time to reach a correct diagnosis.

Previously reported compound score included presence of muscle weakness and CTS history as clinical parameters and amplitude of Sensory action potential (SAP), Compound muscular action potential (CMAP) of the median and ulnar nerves, CMAP of the tibial nerve as electrophysiological parameters. Electrophysiological findings in this study showed that ATTRv patients, although they had the same disease duration of CIAP patients, had a greater reduction of amplitude of potentials in all nerves with a more frequently absence of potential at lower limbs and reduction at upper limbs.

At the same time, the landscape of mutations and phenotypes of ATTR amyloidosis are very different between countries, which does not allow extrapolating the results from Italian study, and there are no comprehensive epidemiological data on patients with hATTR-PN and CIAP in the Russian Federation.

Therefore, there is a need to conduct a large-scale observational study in the Russian population to obtain information on clinical, electrophysiological and demographic characteristics of patients with hATTR-PN and CIAP. Obtaining the study data will help to identify the patients with axonal polyneuropathy, who deserve TTR gene sequencing, and therefore to allow early treatment and potentially modify disease progression in patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hATTR-PN or CIAP ;
* The diagnosis of hATTR-PN or CIAP was established between the 1st January 2017 and the 1st March 2024;
* Presence of at least 1 month between the date of hATTR-PN or CIAP diagnosis and the date of inclusion;
* Age ≥ 18 years at the time of hATTR-PN or CIAP diagnosis.

Exclusion Criteria:

* The participation in any clinical trial with investigational product from the moment of diagnosis of ATTR PN or CIAP until the end of retrospective follow-up period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This non-interventional multicenter observational study will include 50 adult patients with hATTR-PN and 50 adult patients with CIAP in 8 clinical sites in the Russian Federation. The diagnosis should be established in patients' source medical documentation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
In order to describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Mean age at the hATTR-PN or CIAP diagnosis information will be collected | up to 5 months
In order to describe the baseline demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Proportion of women and men will be collected | up to 5 months
In order to describe the baseline demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Proportion of patients with each race and ethnicity will be collected | up to 5 months
to describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIA, information on Proportion of patients from each federal district of the Russian Federation will be collected | up to 5 months
in order to describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, tha following Anthropometric characteristics will be collected: | up to 5 months
  Mean height (in m and cm), body weight (in kg), BMI (kg/m2)
In order to describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients with underweight will be collected | up to 5 months
  BMI <18,5 kg/m2
in order to describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Proportion of patients with negative lifestyle factors will be collected: | up to 5 months
  1. Proportion of patients with a history of smoking;
  2. Proportion of patients with a history of alcohol abuse
in order to describe the baseline demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Proportion of patients with positive family history in close relatives will be collected | up to 5 months
to describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP, information on Mean (or median) time from the first symptoms of neuropathy to the diagnosis of PN will be collected | up to 5 months
to describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP, Proportion of patients with different firstly suspected etiology of PN will be calculated | up to 5 months
  1. Diabetic;
  2. Alcoholic;
  3. Toxic (toxic agents other than alcohol, e.g. drugs or chemotherapy);
  4. Other Hereditary;
  5. Deficiency (due to vitamin B12, thiamine or pyridoxine deficiency);
  6. Immunological (due to rheumatological, paraneoplastic or celiac disease);
  7. Haematological (paraproteinemic syndromes);
  8. Infective;
  9. Idiopathic;
  10. Other;
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP, information on Mean (or median) time from first PN manifestation/diagnosis to the hATTR-PN or CIAP diagnosis will be collected | up to 5 months
To describe the baseline electrophysiological and clinical characteristics of patients, Proportion of patients with chronic sensory or sensorimotor polyneuropathy and progressive chronic polyneuropathy among patients with CIAP will be calculated | up to 5 months
To describe the baseline clinical characteristics of patients with hATTR-PN and CIAP, Proportion of patients with each result of TTR gene testing will be calculated | up to 5 months
  (positive, negative, not performed); the proportion of patients with each identified mutation in TTR gene in case of positive result
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients with each clinical manifestation will be calculated: | up to 5 months
  1. Sensory symptoms;
  2. Motor symptoms;
  3. CTS (proportion of patients with any CTS in total, as well as proportion of patients with uni- and bilateral CTS);
  4. Biceps tendon rupture;
  5. Autonomic symptoms;
  6. Spinal channel stenosis of the lumbar region;
  7. GI symptoms;
  8. Ocular manifestations;
  9. Cardiac manifestations;
  10. Renal manifestations;
  11. CNS involvement.
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients with each PND score will be calculated | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients with each score by each parameter of neurological examination will be calculated | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Mean point by MRS will be calculated | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Mean point by INCAT scale (total score, arm disability, leg disability) will be collected | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Mean left ventricular ejection fraction (LVEF) will be collected | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information Mean wall thickness of the left ventricular (LV) will be collected | up to 5 months
To describe the baseline electrophysiological characteristics of patients with hATTR-PN and CIAP, information Mean variables based on the results of electrophysiological investigation, including the following (on both extremities) will be collected | up to 5 months
  Compound muscular action potential (CMAP) (mV) of the median, ulnar, tibial and peroneal nerves; (b) (Distal motor latency) DML (ms) of the median, ulnar, tibial and peroneal nerves; (c) (Motor nerve conduction velocity) MNCV (m/s) of the median, ulnar, tibial and peroneal nerves; (d) Sensory action potential (SAP) (μV) of the median, ulnar, peroneal superficial and sural nerves; (e) Sensory nerve conduction velocity (SNCV) (m/s) of the median, ulnar, peroneal superficial and sural nerves
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients with diagnosis of HFpEF will be calculated | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Mean NT-proBNP level will be collected | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information Mean estimated glomerular filtration rate (eGFR) will be collected | up to 5 months
  based on CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Mean urine albumin-to-creatinine ratio (UACR) in a spot urine sample will be collected | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients with a positive paraprotein blood test result will be calculated | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, information on Mean blood pressure (BP) (systolic and diastolic) and Mean heart rate (HR) | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients with each concomitant disease will be calculated | up to 5 months
To describe the baseline electrophysiological, clinical and demographic characteristics of patients with hATTR-PN and CIAP in the Russian Federation, Proportion of patients underwent surgery for CTS to the moment of diagnosis will be calculated | up to 5 months

SECONDARY OUTCOMES:
To arrange a score to select patients with axonal neuropathy who deserve screening for TTR mutation. | Up to 5 months
  In order to achieve secondary objective all above baseline demographic, electrophysiological and clinical characteristics will be compared between groups (hATTR-PN and CIAP arm). The score will be arranged based on the parameters by which a significant difference will be determined based on the results of the comparison.

OTHER OUTCOMES:
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP in the Russian Federation during retrospective follow-up period Mean changes in BMI at visits 2, 3 will be compared to baseline | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with newly diagnosed clinical manifestations will be calculated | during retrospective follow-up period
  at visit 2 (in comparison to baseline) and at visit 3 (in comparison to visit 2)
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period, Proportion of patients with different newly diagnosed clinical manifestations will be calculated | during retrospective follow-up period
  at visit 2 (in comparison to baseline) and at visit 3 (in comparison to visit 2)
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with each PND score at visits 2, 3 will be calculated | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP, Proportion of patients with worsening of PND score at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with hospitalisations (one or more) will be calculated | from the date of diagnosis till the end of retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of different reasons for hospitalisations will be calculated | from the date of diagnosis till the end of retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with death for all causes will be calculated | from the date of diagnosis till the end of retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients during follow-up period Proportion of patients with different causes of death will be calculated | from the date of diagnosis till the end of retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients during retrospective follow-up period Proportion of patients with each score by each parameter of neurological examination at visits 2, 3 will be calculated | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in MRS at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in INCAT scale at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
  (total score, arm disability, leg disability)
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with diagnosis of HFpEF at visits 2, 3 will be calculated | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in LVEF at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in wall thickness of the LV at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
To assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
  Mean changes in CMAP, DML, MNCV of the median, ulnar, tibial and peroneal nerves, SAP and SNCV of the median, ulnar, peroneal superficial and sural nerves
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in NT-proBNP at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in eGFR at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in UACR at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with a positive paraprotein blood test result at visits 2, 3 will be calculated | during retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in BP at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Mean changes in HR at visits 2, 3 compared to baseline will be calculated | during retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with new concomitant diseases will be calculated | from the date of diagnosis till the end of retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with different new concomitant diseases will be calculated | from the date of diagnosis till the end of retrospective follow-up period
to assess the changes in the clinical and electrophysiological characteristics of patients with hATTR-PN and CIAP during retrospective follow-up period Proportion of patients with presence of CTS surgery will be calculated | from the date of diagnosis till the end of retrospective follow-up period

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg

REFERENCES:
- See also: D8450R00005 Clinical Study Report (CSR) Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8450R00005&attachmentIdentifier=4a91e694-1643-428d-a946-55f53b8ee7e2&fileName=D8450R00005__Clinical_Study_Report_(CSR)_Synopsis_Redacted.pdf&versionIdentifier=